CLINICAL TRIAL: NCT05709470
Title: Mind the Heart - Mental Health in Children and Adolescents With Congenital Heart Defects in Denmark
Brief Title: Mind the Heart - Mental Health in Children and Adolescents With Congenital Heart Defects
Acronym: Mind the Heart
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Heart Foundation (Other); The Danish DAWBA Center (Unknown); Aalborg University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Sara Hirani Lau-Jensen, Principal Investigater, Rigshospitalet, Denmark
Other Study IDs: P-2021-339
Record Dates: First submitted 2023-01-11; First posted 2023-02-02 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Heart Defects, Congenital; Mental Health Issue
Keywords: Heart Defects, Congenital; Mental Health; Child; Adolescent; Surveys; Questionnaires; Psychiatry
MeSH Terms: conditions — Heart Defects, Congenital; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children and adolescents with congenital heart defects: Children and adolescents between 5-17 years of age, born with a congenital heart defect, living in Denmark at the inclusion time.
  Participants are found though the Danish registries by a diagnosis of congenital heart defect. The diagnosis of Congenital Heart Defect must be given at one of the four University Hospitals in Denmark. These criteria are applied to ensure the validity of the diagnoses.
  Data will be analysed and grouped based on CHD subgroups and as a whole CHD group.
  Interventions: Other: No-intervention

INTERVENTIONS:
Other: No-intervention — Observational cross-sectional study design with no intervention

SUMMARY:
The aim of the Mind the Heart study is to document the feasibility of an online parent/child administered screening model for mental disorders (MDs) in Danish children and adolescents with congenital heart disease (CHD). As MDs in children and adolescents with chronic somatic health issues are frequently underdiagnosed and undertreated, we further aim to develop a website with evidence based information on mental health in children and adolescents with CHD in order to promote knowledge and awareness among families and health professionals across sectors.

DETAILED DESCRIPTION:
Background:

CHD affects approximately 6-10 children per 1000 live births. Innovations in somatic treatment during the last 50 years have increased survival in children with CHD, but also showed a higher risk of cognitive disabilities and MDs like depression, ADHD and autism in children and adolescents with CHD compared to the general population. Untreated childhood MDs may have serious implications for the child's social and academic functioning, quality of life, future health and employment.

Methods:

Danish children and adolescents diagnosed with CHD (N ~ 4800) will be identified through Danish national registries. Parents to eligible children and adolescents will complete bespoke online questionnaires on sociodemographic factors and received psychological support for their children.

Our initial plan was to use the SDQ and DAWBA set-up for the entire CHD group, but based on the low participation rates in the first two CHD groups (the Fontans and ASDs) the set-up was simplified.

The set-up we used is as follows:

Set-up for Fontan and Atrial Septal Defects:

Parents and children ≥ 11 years will complete the internet based Strength and Difficulties Questionnaires (SDQ) and the Development and Wellbeing Assessment (DAWBA). The DAWBA data will be rated by trained clinicians for a possible, probably or no specific psychiatric diagnosis. A summarising report of the results from the DAWBA will be provided to the families within 3 months. Parents will be asked to complete a feasibility questionnaire on the screening procedure, including if they think it would be beneficial to adopt such a procedure in typical clinical practice. The feasibility of the entire online screening procedure will be evaluated.

Set-up for other CHD sub-types:

Parents to children and adolescents will complete the internet based Strength and Difficulties Questionnaire (SDQ). Using the predictive algorithms the probabality of any psychiatric disorder is categorised as either possible, probable or unlikely. Unmet mental health needs will be evaluated.

Emotional and behavioral symptoms and unmet mental health needs will be evaluated in different CHD subtypes separately and across subtypes.

In collaboration with families and cross-sectoral health care providers, a website will be developed. User needs will be identified through semi-structured interviews with representative end users, and the written content will be developed based on a systematic review of the scientific literature, including systematic reviews and meta-analysis, that either illuminates aetiological and maintaining factors for MDs in children and adolescents with CHD, or describes and tests various interventions, and a review of existing information material and management guidelines. The website will be hosted at Rigshospitalet. End user satisfaction will be evaluated through a bespoke questionnaire combined with the System Usability Scale.

The semi-structured interviews with the parents to children and adolescents with CHD and concurrent MDs will further be used for a qualitative study to explore their lived experiences of these issues (Linking Heart and Mind, described elsewhere (https://osf.io/93nb6)).

ELIGIBILITY:
Inclusion Criteria:

* Born with a Congenital Heart Defect
* Age 5-17y
* (Living in Denmark)

Exclusion Criteria:

* Younger than 5years of age
* Older than 17years of age
* Lacking sufficient Danish language skills to answer the questionnaire

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population will be selected though the Danish registries by age and diagnosis of a congenital heart defect (clinical cohort).
Sampling Method: Non-Probability Sample
Enrollment: 4800 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychiatric diagnosis | Day 1
  Number of participants fulfilling the ICD-10/DSM-5 criteria for a psychiatric diagnosis based on the DAWBA.
Emotional and behavioral difficulties | Day 1
  SDQ results will be compared to Danish normative data.

SECONDARY OUTCOMES:
Feasibilty | Day 1
  Feasibilty will be evaluated based on participation rate and acceptability of the screening procedure.
Unmet mental health needs | Day 1
  Mental health service access and unment support needs are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke E Hjortdal, M.D, PhD, professor, Study Director — University of Copenhagen
Locations (1):
- Department of cardiothoracic surgery, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because of the sensitive nature of the data referring to children's psychological profile.